CLINICAL TRIAL: NCT06285071
Title: A Multi-centre, Open-label, Single-arm, Non-interventional Post-marketing Study to Investigate Safety and Clinical Parameters of Alhemo® Under Routine Clinical Practice in Japan
Brief Title: Post-Marketing Surveillance (All Case Surveillance) on Treatment With Alhemo® in Patients With Haemophilia A or Haemophilia B With Inhibitors
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7415-7557; U1111-1274-4740 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — concizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Concizumab: Participants with haemophilia A or haemophilia B with inhibitors will be treated with commercially available Alhemo (Concizumab) according to routine clinical practice at the discretion of the treating physician. Recruitment will be completed after 4.5 years from the launch of Concizumab. The observation period for each participant is 2 years. Total duration of this study is about 6.5 years.
  Interventions: Drug: Concizumab

INTERVENTIONS:
Drug: Concizumab — Participants will be treated with commercially available Alhemo (Concizumab) according to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available Concizumab has been made by the participant/ legally acceptable representative (LAR) and the treating physician before and independently from the decision to include the participant in this study.
  Other Names: Alhemo

SUMMARY:
The purpose of the study is to investigate the safety and effectiveness of Alhemo® in all participants under real-world clinical practice in Japan. Participants will get Alhemo® as prescribed by the study doctor. The study will last for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to initiate treatment with commercially available Alhemo® has been made by the patient/LAR and the treating physician before and independently from the decision to include the patient in this study
* Male or female patients, regardless of age
* Diagnosis with HAwI/HBwI

Exclusion Criteria:

- Previous participation in this study. Participation is defined as having given informed consent in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with haemophilia A or haemophilia B with inhibitors will be treated with commercially available concizumab according to routine clinical practice at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse reaction (AR) | From baseline (week 0) to end of study (week 104)
  Measured as count of ARs.

SECONDARY OUTCOMES:
Number of serious adverse reaction (SAR) | From baseline (week 0) to end of study (week 104)
  Measured as count of SARs.
Number of serious adverse event (SAE) | From baseline (week 0) to end of study (week 104)
  Measured as count of SAEs.
Number of thromboembolic adverse event (AE) | From baseline (week 0) to end of study (week 104)
  Measured as count of thromboembolic AEs.
Number of shock/anaphylaxis AE | From baseline (week 0) to end of study (week 104)
  Measured as count of shock/anaphylaxis AEs.
Number of treated spontaneous and traumatic bleeding episodes | From baseline (week 0) to end of study (week 104)
  Measured as count of bleeding episodes.
Number of treated spontaneous and traumatic target joint bleeding episodes | From baseline (week 0) to end of study (week 104)
  Measured as count of bleeding episodes.
Number of all treatment requiring bleeding episode | From baseline (week 0) to end of study (week 104)
  Measured as count of bleeding episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (7):
- Japan (7):
  - Novo Nordisk Investigational Site, Toshima City, Tokyo
  - Mutsu general hospital, Aomori
  - Kyushu university hospital_Pediatrics, Fukuoka
  - Sapporo Tokushukai Hospital_Pediatrics, Hokkaido
  - Kagoshima City Hospital, Kagoshima
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Tokyo Medical University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com